CLINICAL TRIAL: NCT05476380
Title: Neoadjuvant Therapy of Camrelizumab Combined With Chemotherapy for Resectable Locally Advanced Esophageal Squamous Cell Carcinoma: a Single-arm, Phase II Clinical Study
Brief Title: Neoadjuvant Therapy of Camrelizumab Combined With Chemotherapy for Resectable Locally Advanced Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-OBU-TJ-BB-EC-II-00
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2021-12

CONDITIONS: Esophageal Carcinoma
Keywords: Esophageal Carcinoma; Camrelizumab; Neoadjuvant therapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — camrelizumab; Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CCNT-ESCC (Experimental): This study is a single-arm, open-label, exploratory clinical study, the main purpose of which is to evaluate the efficacy and safety of neoadjuvant treatment of camrelizumab combined with chemotherapy for resectable locally advanced esophageal squamous cell carcinoma.
  After screening, subjects who meet the requirements for entry and exclusion signed the informed consent, received neoadjuvant treatment of carrelizumab combined with combined with chemotherapy.The patient will receive three cycles of treatment of camrelizumab(200 mg, IV., d1, q3w), paclitaxel(175 mg/m2,continuous IV., d1, 24h q3w), cisplatin(75 mg/m2, iv., d1,q3w).Patients who are assessed as being able to undergo surgical resection receive elective resection surgery,and the maintenance treatment of postoperative patients implements individualized treatment.
  Interventions: Drug: camrelizumab

INTERVENTIONS:
Drug: camrelizumab — Camrelizumab:200 mg, IV., d1, q3w; Paclitaxel:175 mg/m2,continuous IV., d1, 24h q3w; Cisplatin:75 mg/m2, iv., d1,q3w
  Other Names: Paclitaxel; Cisplatin

SUMMARY:
To evaluate the efficacy and safety of neoadjuvant therapy of camrelizumab combined with chemotherapy for resectable locally advanced esophageal squamous cell carcinoma

DETAILED DESCRIPTION:
This study is a single-arm, open-label, exploratory clinical study, the main purpose of which is to evaluate the efficacy and safety of neoadjuvant treatment of camrelizumab combined with chemotherapy for resectable locally advanced esophageal squamous cell carcinoma.

The patient will receive three cycles of treatment of camrelizumab(200 mg, IV., d1, q3w), paclitaxel(175 mg/m2,continuous IV., d1, 24h q3w), cisplatin(75 mg/m2, iv., d1,q3w).Patients who are assessed as being able to undergo surgical resection receive elective resection surgery,and the maintenance treatment of postoperative patients implements individualized treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1) Sign the written informed consent before joining the group;
* 2) Age 18-70 years old, both male and female
* 3) T3N+M0 patients with resectable esophageal squamous cell carcinoma confirmed by pathology and imaging（AJCC/UICC eighth edition TNM staging of esophageal cancer）
* 4) Evaluation of patients with locally advanced surgical resection before treatment
* 5) There are measurable lesions that meet the RECIST v1.1 criteria for evaluation;
* 6) ECOG PS score: 0 to 1;
* 7) The expected survival period is greater than 6 months;
* 8) It is allowed to take blood samples and postoperative pathological sections;
* 9) The function of vital organs meets the following requirements (excluding the use of any blood components and cell growth factors within 14 days):

Blood routine:

* Neutrophil ≥1.5*109/L
* Platelet count≥100*109/L
* Hemoglobin ≥ 90g/L;

Liver and kidney function:

* Serum creatinine (SCr) ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance ≥ 50 ml/min (Cockcroft-Gault formula);
* Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≤ 2.5 times the upper limit of normal (ULN); urine protein < 2+; if urine protein ≥ 2+, 24-hour urine protein quantification must show protein ≤ 1 g;
* 10) Normal coagulation function, no active bleeding and thrombotic disease

  1. International Standardized Ratio INR≤1.5×ULN;
  2. Partial thromboplastin time APTT≤1.5×ULN;
  3. Prothrombin time PT≤1.5ULN;
* 11) Non-surgical sterilization or female patients of childbearing age need to use a medically approved contraceptive method (such as an intrauterine device, contraceptives or condoms) during the study treatment period and within 3 months after the end of the study treatment period;Non-surgically sterilized female patients of childbearing age must have a negative serum or urine HCG test within 7 days prior to study enrollment; and must be non-lactating;Non-surgical sterilization or male patients of childbearing age need to agree to use a medically approved contraceptive method with their spouse during the study treatment period and within 3 months after the end of the study treatment period.
* 12）The subjects voluntarily joined the study, with good compliance, and cooperated with safety and survival follow-up

Exclusion Criteria:

* 1) Previously received radiotherapy, chemotherapy, hormone therapy, surgery or molecular targeted therapy;
* 2) Patients with distant metastasis confirmed by imaging;
* 3) The subject has suffered from other malignant tumors in the past or at the same time (except for cured skin basal cell carcinoma and cervical carcinoma in situ);
* 4) Previous treatment with camrelizumab or other PD-1/PD-L1 therapy; known subjects had previous treatment with macromolecular protein preparations, or known treatment with any camrelizumab, paclitaxel or platinum Allergic to ingredients;
* 5) The subject has any active autoimmune disease or has a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis , nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or complete remission of asthma in childhood without any intervention in adulthood can be included; subjects with asthma requiring bronchodilator medical intervention are not included );
* 6) The subject is using immunosuppressive, or systemic, or absorbable local hormone therapy to achieve the purpose of immunosuppression (dose > 10mg/day prednisone or other equivalent hormones), and within 2 weeks before enrollment is still in use;
* 7) Ascites or pleural effusion with clinical symptoms requires therapeutic puncture or drainage;
* 8) There are clinical symptoms or diseases of the heart that cannot be well controlled, such as: (1) NYHA grade 2 or higher heart failure (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
* 9) Abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg>2g/L), with bleeding tendency or receiving thrombolytic or anticoagulation therapy;
* 10) The patient currently (within 3 months) has esophageal varices, active gastric and duodenal ulcers, ulcerative colitis, portal hypertension and other gastrointestinal diseases, or the unresectable tumor has active bleeding, or the investigator determines other conditions that may cause gastrointestinal bleeding and perforation;
* 11) Past or current severe bleeding (bleeding >30 ml within 3 months), hemoptysis (>5 ml fresh blood within 4 weeks), or thromboembolic events (including stroke events and/or transient cerebral insufficiency) within 12 months blood attack);
* 12) The subject has active infection or unexplained fever >38.5 degrees during the screening period and before the first administration (subject to the investigator's judgment, the subject's fever due to tumor can be enrolled);
* 13) Abdominal fistula, gastrointestinal perforation or abdominal abscess occurred less than 4 weeks before study medication;
* 14) Patients with past and current objective evidence of a history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severely impaired lung function, etc.;
* 15) Subjects with congenital or acquired immunodeficiency, such as HIV infection, or active hepatitis (transaminase does not meet the inclusion criteria, hepatitis B reference: HBV DNA ≥ 1000 IU/ml; hepatitis C reference: HCV RNA ≥ 103 IU/ml); Chronic hepatitis B virus carriers, HBV DNA < 2000 IU/ml, must receive antiviral therapy during the trial period before they can be enrolled;
* 16) The subject is participating in other clinical studies or less than 1 month after the end of the previous clinical study; the subject may receive other systemic anti-tumor therapy during the study;
* 17) Less than 4 weeks before the study medication or may be vaccinated with live vaccines during the study period;
* 18) The subject is known to have a history of psychotropic substance abuse, alcohol or drug abuse;
* 19）The researcher believes that it should be excluded from this study. For example, according to the researcher's judgment, the subjects have other factors that may cause the study to be terminated midway. For example, other serious diseases (including mental diseases) require concomitant treatment. Abnormal laboratory tests, accompanied by family or social factors, will affect the safety of subjects, or the collection of data and samples.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
pCR | within 28 working days after operation
  pathological complete response rate

SECONDARY OUTCOMES:
1year DFS rate | Refers to the time from initiation to tumor recurrence or death from any cause (up to approximately 1 year)
  Disease-free survival in 1 year
Postoperative complication rate | within 28 working days after operation
  Postoperative complication rate
R0 resection rate | within 28 working days after operation
  the complete resection rate of all tumor under microscope
DFS | Refers to the time from initiation to tumor recurrence or death from any cause (up to approximately 3 years)
  Disease-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No